CLINICAL TRIAL: NCT04175704
Title: A Phase I, Randomized, Single-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of UB-221 as an Add-on Therapy in Patients With Chronic Spontaneous Urticaria
Brief Title: Evaluating the Safety and Tolerability and Determining the PK and PD of Single Dose UB-221 in Chronic Spontaneous Urticaria
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: United BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBP-A115-IgE
Record Dates: First submitted 2019-11-12; First posted 2019-11-25 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Chronic Idiopathic Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Other): 0.2 mg/kg UB-221 or placebo
  Interventions: Drug: UB-221
- Cohort2 (Other): 0.6 mg/kg UB-221 or placebo
  Interventions: Drug: UB-221
- Cohort 3 (Other): 2 mg/kg UB-221 or placebo
  Interventions: Drug: UB-221
- Cohort 4 (Other): 6 mg/kg UB-221 or placebo
  Interventions: Drug: UB-221

INTERVENTIONS:
Drug: UB-221 — Name: UB-221 Active ingredient: Anti-IgE monoclonal antibody Dosage form: UB-221 drug product is presented as a sterile liquid for intravenous (IV) infusion. Each vial contains 75 mg/mL UB-221 in 1.12 mL of buffered solution
  Other Names: recombinant anti-IgE humanized IgG1 monoclonal antibody

SUMMARY:
The study is to evaluate the profiles of safety, tolerability, pharmacokinetics, and pharmacodynamics of UB-221. In this study, safety profile of UB-221 and maximum tolerated dose (MTD) is to be investigated using sentinel dosing strategy. The starting dose of 0.2 mg/kg is selected based on the evaluation and comparison of various approaches including NOAEL, MABEL (minimum anticipated biological effect level), and experiences from other anti-IgE mAb drugs in development.

DETAILED DESCRIPTION:
This is a phase I, randomized, single-blind, placebo-controlled, parallel group, single ascending dose study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of a single dose of UB-221 as an add-on therapy in chronic spontaneous urticaria (CSU) subjects who fail to respond to the first line H1-antihistamine treatment. Only the qualified subjects will be blinded to receive treatment. Each subject will receive only one dose of UB-221 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 years
* Subjects who are able and willing to provide the informed consent
* Subjects diagnosed with chronic spontaneous urticaria (CSU) for more than six weeks prior to the screening visit as confirmed by investigators based on medical history.

Exclusion Criteria:

* History of significant diseases (other than CSU) or major clinical conditions by the investigator's judgment, such as auto-immune disease or psychiatric and behavioral conditions from which the investigator considers the subject not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety (Adverse event (AE)/ serious adverse event (SAE)) of UB-221 in CSU patients | 99 days
  1.Adverse event (AE)/ serious adverse event (SAE) reporting: from treatment to EOS